CLINICAL TRIAL: NCT04921761
Title: Dural Puncture Epidural Technique Versus Conventional Epidural Technique During Vaginal Surgeries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There is a duplicate study registered. The trial registration and later updates will be in NCT04933500. That is the record that will be updated.
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Dural Puncture
Record Dates: First submitted 2021-06-05; First posted 2021-06-10 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Dural Puncture Epidural Technique

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): Women who received the conventional epidural technique (group A). Intervention: Procedure: Conventional epidural
  Interventions: Procedure: Conventional epidural
- Group B (Active Comparator): Women who received the dural puncture epidural technique (group B). Intervention: Procedure: Dural puncture epidural
  Interventions: Procedure: Dural puncture epidural

INTERVENTIONS:
Procedure: Conventional epidural — In this group, a 20-gauge multi-orifice catheter was threaded through the cephalic-directed tip of the epidural needle 5 cm into the epidural space.
  Arms: Group A
Procedure: Dural puncture epidural — In this group, the dura was punctured by 25G Whitacre needle. After confirmation of CSF flow, the needle was removed and the epidural catheter was threaded.
  Arms: Group B

SUMMARY:
The study aims to evaluate whether the dural puncture epidural technique (group B) improves sacral block anesthesia during vaginal surgeries compared with the conventional epidural technique (group A).

ELIGIBILITY:
Inclusion Criteria:

Age (25- 55) years. Height (150 -170) cm.

Exclusion Criteria:

Patient refusal. Hypersensitivity to local anesthetic drugs. Bleeding disorders and coagulopathy. Severe mitral or aortic stenosis. Local or systemic sepsis. Uncooperative patients. Sever spinal deformity. Blood or CSF in the epidural catheter during the procedure. Failure of the block and need for general anesthesia.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Time of onset of anesthesia to T10 | During surgery
Time for complete motor block | During surgery
Time for first rescue analgesia will be required during surgery | During surgery